CLINICAL TRIAL: NCT00558636
Title: A Randomized Controlled Trial Comparing Safety and Efficacy of Carboplatin and Paclitaxel Plus or Minus Sorafenib (BAY43-9006) in Chemonaive Patients With Stage IIIB-IV Non-Small Cell Lung Cancer (NSCLC)
Brief Title: A Trial Comparing Safety and Efficacy of Carboplatin and Paclitaxel Plus or Minus Sorafenib (BAY43-9006) in Chemonaive Patients With Stage IIIB-IV Non-Small Cell Lung Cancer (NSCLC)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Terminated early when the results from Study NCT00300885 showed an overall lack of efficacy in NSCLC and increased mortality in subjects with squamous subtype.
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 12621
Record Dates: First submitted 2007-11-09; First posted 2007-11-15 (Estimated); Results first posted 2010-10-20 (Estimated); Last update posted 2013-12-27 (Estimated); Status verified 2013-12

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Sorafenib; Paclitaxel; Carboplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sorafenib + Paclitaxel + Carboplatin (Experimental): Chemotherapy plus Multi Kinase Inhibitor: Sorafenib Group - Sorafenib (Nexavar, BAY43-9006), [400 mg, (2 tablets x 200 mg each) orally, twice daily] on Study Days 2-19 and paclitaxel (175 mg/m^2, intravenous (IV), over 2.5 to 4 hours) and carboplatin (area under the curve (AUC) =5, IV for 15 to 60 minutes) on Study Day 1. The cycle duration will be 21 days.
  Interventions: Drug: Sorafenib + Paclitaxel + Carboplatin
- Placebo + Paclitaxel + Carboplatin (Placebo Comparator): Chemotherapy + Placebo: Placebo Group - Placebo (2 tablets twice daily, orally) on Study Days 2-19 and paclitaxel (175 mg/m^2 IV, over 2.5 to 4 hours) and carboplatin (AUC=5 IV, for 15 to 60 minutes) on Study Day 1. The cycle duration will be 21 days
  Interventions: Drug: Placebo + Paclitaxel + Carboplatin

INTERVENTIONS:
Drug: Sorafenib + Paclitaxel + Carboplatin — Chemotherapy plus Multi Kinase Inhibitor: Sorafenib Group - Sorafenib (Nexavar, BAY43-9006), [400 mg, (2 tablets x 200 mg each) orally, twice daily] on Study Days 2-19 and paclitaxel (175 mg/m^2, intravenous (IV), over 2.5 to 4 hours) and carboplatin (area under the curve (AUC) =5, IV for 15 to 60 minutes) on Study Day 1. The cycle duration will be 21 days.
  Arms: Sorafenib + Paclitaxel + Carboplatin
Drug: Placebo + Paclitaxel + Carboplatin — Chemotherapy + Placebo: Placebo Group - Placebo (2 tablets twice daily, orally) on Study Days 2-19 and paclitaxel (175 mg/m^2 IV, over 2.5 to 4 hours) and carboplatin (AUC=5 IV, for 15 to 60 minutes) on Study Day 1. The cycle duration will be 21 days
  Arms: Placebo + Paclitaxel + Carboplatin

SUMMARY:
The purpose of this study conducted in Asia-Pacific was to evaluate the efficacy and safety of Sorafenib in combination with paclitaxel and carboplatin versus placebo in combination with paclitaxel and carboplatin for chemonaive patients with unresectable stage IIIB (with effusion) or stage IV NSCLC. However, as indicated below, the study was terminated prematurely when the results from Study 11961 (NCT00300885), an earlier Phase 3 study of similar design in subjects with advanced NSCLC, showed an overall lack of efficacy and increased mortality in subjects with squamous subtype. The data available is presented as descriptive analyses, due to the limitations of implementing the statistical analysis plan.

DETAILED DESCRIPTION:
The study was terminated early when the results from Study 11961 (NCT00300885), an earlier Phase 3 study evaluating the effects of Sorafenib in combination with paclitaxel and carboplatin in subjects with advanced NSCLC, showed an overall lack of efficacy of Sorafenib in combination with paclitaxel and carboplatin in NSCLC and increased mortality in subjects with squamous subtype.

ELIGIBILITY:
Inclusion Criteria:

* Stage IIIB (with cytologically confirmed malignant pleural or pericardial effusion) or Stage IV histological or cytological confirmation of NSCLC (thoracentesis or pericardiocentesis is not necessary if a biopsy of the original tumor is available to confirm diagnosis of NSCLC)
* Patients must have measurable disease according to response evaluation criteria in solid tumors (RECIST) criteria
* Prior local radiotherapy is allowed if it is completed at least 3 weeks prior to the first dose of study drug, but the lesion which undergo RECIST assessment should not be in the field of the prior radiation
* Prior surgery is allowed if it is performed at least 4 weeks prior to the first dose of study drug
* 18 years and above
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Life expectancy of at least 12 weeks
* Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements to be conducted within 7 days prior to start of first dose:
* Hemoglobin 9.0 g/dl
* Absolute neutrophil count (ANC) 1,500/mm3
* Platelet count 100,000/mm3
* Total bilirubin < 1.5 times the upper limit of normal
* alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 2.5 x upper limit of normal (< 5 x upper limit of normal for patients with liver involvement)
* international normalized ratio (INR) < 1.5 and activated or adjusted partial thromboplastin time (APTT) within normal limits (1.2 times the lower limit of normal (LLN) to 1.2 times the upper limit of normal (ULN))
* Creatinine </= 1.5 times the upper limit of normal
* Ability to understand and the willingness to sign a written informed consent. A signed informed consent must be obtained prior to any study specific procedures

Exclusion Criteria:

* Any prior systemic anticancer therapy including cytotoxic therapy, targeted agents, experimental therapy, adjuvant, or neo-adjuvant therapy for any current or prior diagnosis of NSCLC
* Cardiac disease: Congestive heart failure > class II New York Heart Association (NYHA). Patients must not have unstable angina (anginal symptoms at rest) or new-onset angina (began within the last 3 months) or myocardial infarction within the past 6 months
* Known brain metastasis. Patients with neurological symptoms should undergo at Computed Tomography (CT) scan/Magnetic Resonance Imaging (MRI) of the brain to exclude brain metastasis
* Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
* Uncontrolled hypertension defined as systolic blood pressure > 150 mm Hg or diastolic pressure > 90 mm Hg, despite optimal medical management
* Known human immunodeficiency virus (HIV) infection
* Active clinically serious infections > Common Terminology Criteria for Adverse Events (CTCAE) Grade 2
* Thrombotic or embolic events such as cerebrovascular accident including transient ischemic attacks within the past 6 months
* Pulmonary hemorrhage/bleeding event > CTCAE Grade 2 within 4 weeks of first dose of study drug
* Any other hemorrhage/bleeding event > CTCAE Grade 3 within 4 weeks of first dose of study drug
* Serious, non-healing wound, ulcer, or bone fracture
* Evidence or history of bleeding diathesis or coagulopathy
* Major surgery, open biopsy or significant traumatic injury within 4 weeks of first dose of study drug
* Therapeutic anticoagulation with vitamin K antagonists such as warfarin, or with heparins or heparinoids. Low dose warfarin (1 mg daily, oral) is permitted if the INR remains < 1.5. Low-dose aspirin is permitted
* Known or suspected allergy to sorafenib or any agent given in the course of this trial
* Cancer other than NSCLC within 5 years prior to start of study treatment, EXCEPT cervical cancer in-situ, treated basal cell carcinoma, or superficial bladder tumors
* Concurrent cancer that is distinct in primary site or histology from NSCLC
* Substance abuse, medical, psychological or social conditions that may interfere with the patients participation in the study or evaluation of the study results
* Any condition that impairs patients ability to swallow whole pills
* Any malabsorption condition
* Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of treatment
* Women of childbearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation, including the 30 days period after last study drug dosing. The investigator should advise the patient how to achieve an adequate contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2007-09; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (15):
- China (7):
  - Guangzhou, Guangdong
  - Shatin, Hong Kong
  - Nanjing, Jiangsu
  - Hangzhou, Zhejiang
  - Beijing
  - Chongqing
  - Shanghai
- India (2):
  - Mumbai, Maharashtra
  - New Delhi
- Singapore, Singapore
- South Korea (2):
  - Gyeonggi-do
  - Seoul
- Taiwan (2):
  - Taipei, Taiwan
  - Changhua
- Bangkok, Bangkok, Thailand

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 23 Sep 2007 to 12 May 2008 (first subject's first visit to last subject's last visit) at 15 centers in 4 countries: China (9), Singapore (2), Thailand (2), and Taiwan (2). The study was terminated prematurely after about 5 months of recruitment and before the planned 230 progression free survival (PFS) events occurred.
Pre-assignment Details: At the time of study termination, 91 (out of 108 screened subjects) of the planned 294 subjects had been screened and randomized. All 91 randomized subjects received at least 1 dose of study drug and were included in both the intent-to-treat (ITT) and safety analysis populations.
Period: Treatment
Arm/Group | Sorafenib + Paclitaxel + Carboplatin | Placebo + Paclitaxel + Carboplatin
Started | 47 (up to 6 cycles of combination therapy) | 44
Start of Maintenance Monotherapy | 2 (Sorafenib taken as the single agent in the Maintenance Phase) | 2 (Placebo taken as the single agent in the Maintenance Phase)
Completed | 0 (Patients still on treatment did not enter follow-up because the study was prematurely terminated) | 0 (Patients still on treatment did not enter follow-up because the study was prematurely terminated)
Not Completed | 47 | 44
Not completed — Adverse Event | 9 | 2
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Premature termination of the study | 35 | 37
Not completed — Disease progression | 1 | 5
Period: Follow-up
Arm/Group | Sorafenib + Paclitaxel + Carboplatin | Placebo + Paclitaxel + Carboplatin
Started | 12 (12 subjects entered Follow-up phase before they completed the treatment phase) | 7 (7 subjects entered Follow-up phase before they completed the treatment phase)
Completed | 0 (Study was prematurely terminated) | 0 (Study was prematurely terminated)
Not Completed | 12 | 7
Not completed — Premature termination of the study | 12 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sorafenib + Paclitaxel + Carboplatin | Placebo + Paclitaxel + Carboplatin | Total
Number analyzed (Participants) | 47 | 44 | 91
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 38 | 32 | 70
  >=65 years | 9 | 12 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.2 (9.3) | 55.4 (12.6) | 55.8 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 14 | 34
  Male | 27 | 30 | 57
Eastern Cooperative Oncology Group (ECOG) performance status [Number; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status is a scale that measures how cancer affects a patient. The scale ranges from 0 (fully active) to 5 (dead). Subjects entering this study must have had an ECOG score of 0 or 1(restricted in physically strenuous activity but ambulatory).
  Participants
    Grade 0: Fully active | 8 | 5 | 13
    Grade 1: Restricted strenuous activity, ambulatory | 39 | 39 | 78
Geographic region [Number; unit: Participants] — Subjects in the study were stratified as to whether they were from China or not from China.
  Participants
    China | 35 | 36 | 71
    Non-China | 12 | 8 | 20
Histology [Number; unit: Participants] — Subjects in the study were stratified by the histology of their non-small cell lung cancer into non-squamous vs squamous.
  Participants
    Squamous cell (epidermoid) carcinoma | 13 | 14 | 27
    Other | 33 | 30 | 63
    Missing histology | 1 | 0 | 1
Stage at study entry [Number; unit: Participants] — Subjects in the study were stratified by the stage of their disease: Stage IIIB (with cytologically confirmed malignant pleural or pericardial effusion) or Stage IV histological or cytological confirmation of Non-Small Cell Lung Cancer (NSCLC).
  Participants
    Missing | 3 | 1 | 4
    Stage IIIB | 7 | 3 | 10
    Stage IV | 37 | 40 | 77

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Progression free survival (PFS) is the time (days) from date of randomization to date of first observed disease progression (radiological or clinical, whichever was earlier) or death due to any cause, if death occurred before progression was documented. Since the study was terminated early and 89% of subjects' data were censored, only the number of PFS events (Failed [progressed or died before progression]) is reported, not the usual measure "number of days".
Time Frame: Up to 5 months after randomization of the first patient
Population: It was intended to include all randomized subjects (the intent to treat (ITT) population) in the analysis. Since 89% of subjects were censored, PFS could not be calculated. The number of subjects who Failed (progressed or died before progression) or were Censored are reported.
Measure: Number; unit: Participants
Arm/Group | Sorafenib + Paclitaxel + Carboplatin | Placebo + Paclitaxel + Carboplatin
Number analyzed (Participants) | 47 | 44
Participants
  Failed (progressed or died before progression) | 5 | 5
  Censored | 42 | 39

2. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is the number of days from the date of randomization to the date of death due to any cause. Subjects alive at the time of analysis were censored at their last date of follow-up. Since the study was terminated early and 89% of subjects' data were censored, only the number of subjects who Failed (died) or were Censored is reported, not the usual measure "number of days".
Time Frame: Up to 5 months after randomization of the first patient
Population: All randomized subjects (the intent to treat (ITT) population) were included in the analysis. Since 89% of subjects were censored, OS could not be calculated. The number of subjects who Failed (died) or were Censored are reported.
Measure: Number; unit: Participants
Arm/Group | Sorafenib + Paclitaxel + Carboplatin | Placebo + Paclitaxel + Carboplatin
Number analyzed (Participants) | 47 | 44
Participants
  Failed (died) | 4 | 1
  Censored | 43 | 43

3. Secondary Outcome: Best Tumor Response (Number of Responses Per Category) According to Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Complete response (CR): Disappearance of all target lesions (TL). Partial response (PR): At least 30% decrease in sum of the largest diameter (LD) of TLs, taking baseline sum as reference. Stable disease (SD): No change in tumor size. Progressive disease (PD): At least a 20% increase in the sum of the LD of TLs, taking as reference the smallest sum LD recorded since treatment started, or the appearance of 1 or more new lesions.
Time Frame: Best tumor response assessed every 6 weeks by investigator during treatment up to 5 months after randomization of the first patient.
Population: All randomized subjects (the intent to treat (ITT) population) were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Sorafenib + Paclitaxel + Carboplatin | Placebo + Paclitaxel + Carboplatin
Number analyzed (Participants) | 47 | 44
Participants
  Complete repsonse (CR) | 0 | 0
  Partial response (PR) | 4 | 0
  Stable disease (SD) | 18 | 28
  Progressive disease (PD) | 1 | 1
  not evaluated | 24 | 15

4. Secondary Outcome: Duration of Response
Description: Duration of response (PR or better) was defined as the time from the first documented objective PR or CR, whichever was noted earlier, to disease progression or death (if death occurred before progression was documented). Since only 4 subjects had a response, the duration of response was not calculated.
Time Frame: Time from first documented objective response (complete response or partial response) to disease progression or death, or to last tumor assessment if censored, up to 5 months after randomization of the first patient.
Population: All subjects that showed a response. Since only 4 subjects had a response, the data were not analyzed.
Measure: Number; unit: days
Arm/Group | Sorafenib + Paclitaxel + Carboplatin | Placebo + Paclitaxel + Carboplatin
Number analyzed (Participants) | 4 | 0
days
  The first subject who showed a response | 91 |
  The second subject who showed a response | 45 |
  The third subject who showed a response | 46 |
  The fourth subject who showed a response | 53 |

5. Secondary Outcome: Change From Baseline of Lung Cancer Symptoms (LCS) Score Assessed at Each Treatment Cycle (21 Days Per Cycle) Starting With Cycle 2
Description: The LCS is a validated instrument for determining treatment impact on lung symptoms. The LCS consists of 7 questions with 5 responses ranging from "not at all" to "very much". The LCS total score ranges from 0 to 28. Lower scores reflect greater lung cancer symptoms.
Time Frame: Change from baseline of LCS score assessed at each treatment cycle starting with Cycle 2 (Cycles 2, 3, 4, 5, 6, 7; 21 days per cycle) up to 5 months after randomization of the first patient.
Population: Of the 91 randomized subjects in the ITT population, 90 completed the LCS at baseline. Since more than half of the subjects received only 1 or 2 cycles before the trial was stopped, the response rate (number of evaluable subjects completing the questionnaire) decreased from cycle to cycle and makes the results hard to interpret.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sorafenib + Paclitaxel + Carboplatin | Placebo + Paclitaxel + Carboplatin
Number analyzed (Participants) | 47 | 43
units on a scale
  Cycle 2 (N = 31 sorafenib/33 placebo) | 2.8 (10.0) | 1.1 (5.6)
  Cycle 3 (N = 16 sorafenib/23 placebo) | 0.4 (3.6) | 0.2 (13.2)
  Cycle 4 (N = 12 sorafenib/14 placebo) | -0.1 (3.0) | 2.2 (4.2)
  Cycle 5 (N = 7 sorafenib/5 placebo) | 2.4 (2.7) | 3.6 (4.5)
  Cycle 6 (N = 4 sorafenib/3 placebo) | -0.8 (2.9) | 4.3 (8.6)
  Cycle 7 (N = 2 sorafenib/1 placebo) | 3.0 (2.8) | 0 (0)

6. Secondary Outcome: Change From Baseline of Health-Related Quality of Life (HRQoL) Score Assessed at Treatment Cycle 3 and Cycle 5
Description: HRQoL was assessed with the Functional Assessment of Cancer Therapy-Lung (FACT-L) questionnaire, a validated instrument for determining lung cancer HRQoL. The 36-item questionnaire includes 4 domains: Physical, functional, emotional, and social/family well-being, and a lung cancer-specific subscale. The FACT-L total score ranges from 1 to 136. Lower scores demonstrate impaired HRQoL.
Time Frame: Change from baseline of HRQoL score assessed (at treatment Cycle 3 and Cycles 5 [21 days per cycle]) up to 5 months after randomization of the first patient.
Population: Of the 91 randomized subjects in the ITT population, 88 completed the FACT-L at baseline. Since more than half of the subjects received only 1 or 2 cycles before the trial was stopped, the number of subjects who completed the questionnaire after the first cycles was very low, making the results difficult to interpret.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sorafenib + Paclitaxel + Carboplatin | Placebo + Paclitaxel + Carboplatin
Number analyzed (Participants) | 46 | 42
units on a scale
  Cycle 3 (N = 16 sorafenib/21 placebo) | -5.1 (10.6) | 4.6 (19.5)
  Cycle 5 (N = 7 sorafenib/5 placebo) | 0 (9.9) | 11.2 (27.8)

7. Secondary Outcome: Change From Baseline of Health-Related Quality of Life (HRQoL) Score Assessed at Treatment Cycle 7
Description: as for outcome 6
Time Frame: Change from baseline of HRQoL score assessed (at treatment Cycle 7 [21 days per cycle]) up to 5 months after randomization of the first patient.
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Sorafenib + Paclitaxel + Carboplatin | Placebo + Paclitaxel + Carboplatin
Number analyzed (Participants) | 2 | 1
Units on a scale | 13.5 (6.4) | 11.3

ADVERSE EVENTS:
Description: The following acronyms and abbreviations were used in the Results section: Absolute Neutrophil Count (ANC); Not Otherwise Specified (NOS); Alanine aminotransferase (ALT); Gastrointestinal (GI)
Arm/Group | Sorafenib + Paclitaxel + Carboplatin | Placebo + Paclitaxel + Carboplatin
Serious Adverse Events (participants affected / at risk) | 11/47 | 3/44
Other Adverse Events (participants affected / at risk) | 45/47 | 39/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib + Paclitaxel + Carboplatin (N=47) | Placebo + Paclitaxel + Carboplatin (N=44)
Allergic reaction (Immune system disorders) | 0 | 1
Neutrophiles (Blood and lymphatic system disorders) | 1 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2 | 0
Rash/Desquamation (Skin and subcutaneous tissue disorders) | 2 | 0
Febrile Neutropenia (Infections and infestations) | 3 | 0
Infection (documented clinically), Lung (Pneumonia) (Infections and infestations) | 1 | 0
Infection with normal ANC, blood (Infections and infestations) | 1 | 0
Pain, abdomen NOS (General disorders) | 1 | 0
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Thrombosis/Embolism (vascular access) (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib + Paclitaxel + Carboplatin (N=47) | Placebo + Paclitaxel + Carboplatin (N=44)
Hemoglobin (Blood and lymphatic system disorders) | 12 | 5
Leukocytes (Blood and lymphatic system disorders) | 14 | 10
Neutrophils (Blood and lymphatic system disorders) | 31 | 25
Platelets (Blood and lymphatic system disorders) | 18 | 7
Fatigue (General disorders) | 11 | 12
Fever (General disorders) | 13 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 18 | 16
Hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 19 | 2
Rash/Desquamation (Skin and subcutaneous tissue disorders) | 23 | 6
Anorexia (Gastrointestinal disorders) | 6 | 10
Diarrhea (Gastrointestinal disorders) | 14 | 7
Neuropathy: sensory (Nervous system disorders) | 8 | 12
Allergic reaction (Immune system disorders) | 6 | 2
Lymphopenia (Blood and lymphatic system disorders) | 4 | 4
Supraventricular arrhythmia, sinus tachycardia (Cardiac disorders) | 0 | 3
Hypertension (Cardiac disorders) | 8 | 1
Insomnia (General disorders) | 3 | 1
Constipation (Gastrointestinal disorders) | 8 | 8
GI-other (Gastrointestinal disorders) | 3 | 0
Nausea (Gastrointestinal disorders) | 7 | 5
Vomiting (Gastrointestinal disorders) | 7 | 4
ALT (Metabolism and nutrition disorders) | 5 | 3
Hyperglycemia (Metabolism and nutrition disorders) | 6 | 3
Hyperuricemia (Metabolism and nutrition disorders) | 2 | 3
Hypokalemia (Metabolism and nutrition disorders) | 5 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 2 | 4
Hyponatremia (Metabolism and nutrition disorders) | 8 | 4
Hypophosphatemia (Metabolism and nutrition disorders) | 6 | 0
Lipase (Metabolism and nutrition disorders) | 9 | 2
Pain, bone (General disorders) | 3 | 2
Pain, extremity-limb (General disorders) | 2 | 6
Pain, joint (General disorders) | 2 | 7
Pain, muscle (General disorders) | 7 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 3 | 3

LIMITATIONS AND CAVEATS:
Due to early termination of the study, no comparison of treatments was possible. This study also provided limited opportunity to distinguish between Adverse Events associated with sorafenib and events associated with the underlying lung disease.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less